CLINICAL TRIAL: NCT03120286
Title: OVERWEIGHT AND OBESITY ADVERSELY AFFECT IN VITRO FERTILIZATION (IVF) OUTCOMES IN WOMEN WITH POLYCYSTIC OVARY SYNDROME (PCOS)
Brief Title: OVERWEIGHT AND OBESITY ADVERSELY AFFECT IVF OUTCOMES IN WOMEN WITH PCOS
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Saber Thabet Abdalmageed, Principal invistigator, Assiut University
Other Study IDs: BMI
Record Dates: First submitted 2017-04-15; First posted 2017-04-19 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Polycystic Ovary Syndrome IVF
Keywords: OBESITY; In Vitro Fertilization (IVF); Polycystic ovary syndrome (PCOS)
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Overweight and obesity: Women with BMI >25
- Normal weight group: Women with BMI =18-24

SUMMARY:
The effect of overweight and obesity on IVF outcomes is still questionable. The purpose of this study was to determine if overweight/obesity in women with PCOS were associated with an adverse IVF outcome compared to those with normal weight.

Design: Retrospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* All women within the age limit

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is a retrospective study to evaluate the impact of obesity on ivf outcomes.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Live birth rate | On the date of delivery
  Number of live births divided by the number of aspiration cycle

IPD SHARING:
Plan to Share IPD: No